CLINICAL TRIAL: NCT02819661
Title: Difference in the Frequency of Episodes of Respiratory Depression Between Obese (BMI≥30) and Women With Normal BMI Receiving Spinal Anesthesia Combined With Intrathecal Morphine During Elective Caesarean Section
Brief Title: Respiratory Depression in Women With BMI≥30 Underwent Spinal Anesthesia With Intrathecal Morphine in Elective C-section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0202-16-RMB CTIL
Record Dates: First submitted 2016-06-15; First posted 2016-06-30 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Depression
Keywords: Elective Caesarean Section; obese women; BMI≥30; spinal anesthesia combined with intrathecal morphine
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Cesarean Section; Anesthesia, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- women BMI<30 POD 1 (Active Comparator): Pregnant healthy women with BMI<30 receiving spinal anesthesia with intrathecal morphine during elective caesarean section will be monitored by SOMNOTOUCH RESP post operative day 1 after elective cesarean section.
  Interventions: Device: SOMNOTOUCH RESP; Procedure: Caesarean section; Drug: Spinal anesthesia with intrathecal morphine
- women BMI≥30 POD 1 (Active Comparator): Pregnant healthy women with BMI≥30 receiving spinal anesthesia with intrathecal morphine during elective caesarean section will be monitored by SOMNOTOUCH RESP post operative day 1 after elective cesarean section.
  Interventions: Device: SOMNOTOUCH RESP; Procedure: Caesarean section; Drug: Spinal anesthesia with intrathecal morphine
- women BMI<30 POD4 (Active Comparator): Pregnant healthy women with BMI<30 receiving spinal anesthesia with intrathecal morphine during elective caesarean section will be monitored by SOMNOTOUCH RESP post operative day 4 after elective cesarean section.
  Interventions: Device: SOMNOTOUCH RESP; Procedure: Caesarean section; Drug: Spinal anesthesia with intrathecal morphine
- women BMI≥30 POD 4 (Active Comparator): Pregnant healthy women with BMI≥30 receiving spinal anesthesia with intrathecal morphine during elective caesarean section will be monitored by SOMNOTOUCH RESP post operative day 4 after elective cesarean section.
  Interventions: Device: SOMNOTOUCH RESP; Procedure: Caesarean section; Drug: Spinal anesthesia with intrathecal morphine

INTERVENTIONS:
Device: SOMNOTOUCH RESP — Ventilatory effort recorder
Procedure: Caesarean section — Cesarean delivery is defined as the delivery of a fetus through surgical incisions made through the abdominal wall (laparotomy) and the uterine wall (hysterotomy).
Drug: Spinal anesthesia with intrathecal morphine — is a form of regional anaesthesia involving injection of a local anaesthetic into the subarachnoid space
  Other Names: Subarachnoid block with intrathecal morphine; spinal block with intrathecal morphine

SUMMARY:
The study will examine whether there is a difference in the frequencies of respiratory depression among obese women receiving spinal anesthesia combined with opioids compared to women with normal BMI.

If such a risk exists further investigation will be required to establish the proper criteria for the administration of morphine with spinal anesthesia to obese women.

DETAILED DESCRIPTION:
Since 1979, intrathecal morphine combined with spinal anesthesia has been shown to provide effective postoperative analgesia in a variety of surgeries and more specifically in caesarean sections.

The advantages of addition of morphine to spinal analgesia are in prolonged analgesia during the operation and post operatively. In addition the analgesia is provided using a single injection during the time of surgery with no further need for complex and costly instruments like an opioid pump .

The side effects and risks of intrathecal morphine include: nausea, vomiting, pruritus urinary retention and the most severe being respiratory depression (immediate or delayed). The mild side effects were higher postoperatively in patients receiving spinal anesthesia combined with morphine. In a meta-analysis study of different surgeries performed under spinal anesthesia, it has been shown that at low doses (<0.3mg) intrathecal morphine does not increase the rate of respiratory depression. Nonetheless higher doses (>0.3mg) were associated with more incidents of respiratory depression. In another study there was no evidence of respiratory depression following caesarean section under spinal anesthesia combined with morphine. Yet, in a prospective study that reviewed 856 cases of caesarean sections under spinal anesthesia combined with morphine a rate of 8 incidences of respiratory depression were found. In a retrospective study of 1915 cases of women undergoing caesarean section with spinal anesthesia combined with morphine a rate of 0.25% of respiratory depression was reported.

The definition of respiratory depression is the lack of response to hypercapnia and/or hypoxia and it has been shown that intrathecal morphine depresses both responses. The common parameters that are monitored in order to detect respiratory depression include respiratory rate, sedation score, pulse oximetry, high PCo2 levels and the need for naloxone treatment. However, the overall measurement of frequency of respiratory depression postoperatively is variable. Accounting for this variability is the fact that hypercapnia may occur in patients with normal respiratory rate, normal sedation score and normal oxygen saturation. In addition, respiratory depression detected by high levels of PCo2 may be recognized earlier than with other parameters.

The risk factors that were found to be associated with respiratory depression included high BMI, prior opioid use, magnesium infusion and respiratory comorbidities In a study of 856 women 8 of them experienced oxygen desaturation during sleep. All of these women were extremely obese with a prior history of deep snoring.

In this study the investigators would like to examine whether there is a difference in the frequency of episodes of respiratory depression between obese (BMI≥30) and women with normal BMI receiving spinal anesthesia combined with intrathecal morphine during elective caesarean section. In previous studies it was reported that obese and non-obese women do not respond differently to modest doses of spinal anesthesia. Hence in this study the investigators can be certain that the investigators are examining the influence of addition of morphine to the spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy
* Healthy women

Exclusion Criteria:

* Heart diseases
* Autoimmune diseases
* Respiratory diseases

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinical respiratory depression by SOMNOtouchTM device monitoring | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam healthcare campus, Haifa, Isreal, Israel

IPD SHARING:
Plan to Share IPD: No